CLINICAL TRIAL: NCT01319487
Title: A 6-month, Phase II, Double-masked, Multicenter, Randomized, Placebo Controlled, Parallel Group Study to Assess the Safety and Efficacy of Topical Administration of Two Concentrations of FOV2304 (High Dose or Low Dose) for the Treatment of Center-involving Clinically Significant Macular Edema Associated With Diabetic Retinopathy
Brief Title: Safety and Efficacy Study of Topical Administration of FOV2304 (High Dose or Low Dose) for the Treatment of Center-involving Clinically Significant Macular Edema Associated With Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fovea Pharmaceuticals SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FOV2304/CLIN/201/P
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-08

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2304 Eye Drops High Dose (Experimental): 2304 Eye Drops High Dose self-administered in the study eye during the treatment period
  Interventions: Drug: 2304 Eye Drops High Dose
- 2304 Eye Drops Low Dose (Experimental): 2304 Eye Drops Low Dose self-administered in the study eye during the treatment period
  Interventions: Drug: 2304 Eye Drops Low Dose
- Placebo Eye Drops (Placebo Comparator): Placebo Eye Drops self-administered in the study eye during the treatment period
  Interventions: Drug: Placebo Eye Drops

INTERVENTIONS:
Drug: 2304 Eye Drops High Dose — 2304 Eye Drops High Dose self-administered in the study eye during the treatment period
  Arms: 2304 Eye Drops High Dose
Drug: 2304 Eye Drops Low Dose — 2304 Eye Drops Low Dose self-administered in the study eye during the treatment period
  Arms: 2304 Eye Drops Low Dose
Drug: Placebo Eye Drops — Placebo Eye Drops self-administered in the study eye during the treatment period
  Arms: Placebo Eye Drops

SUMMARY:
The purpose of the study is to determine whether concentrations of FOV2304 (high dose or low dose) administered in the eye are more effective than placebo in treating patients with diabetic macular edema, following 12 weeks of treatment.

ELIGIBILITY:
Main inclusion/exclusion criteria are listed below. Others may apply.

Inclusion Criteria:

1. Male or female, at least 18 years of age.
2. Diagnosis of diabetes mellitus
3. Patient must be able to self administer study drug.
4. Clinically significant diabetic macular edema in at least one eye ("study eye") involving the center of the macula:
5. Mild to severe non proliferative diabetic retinopathy (Early Treatment Diabetic Retinopathy Study [ETDRS] grade between 20 and 53).
6. BCVA score ≥ 34 letters and < 80 letters in the study eye.
7. Women of childbearing potential must have a negative urine pregnancy test at Screening and be using two highly effective methods of contraception throughout the study.
8. Male patients with partners of childbearing potential must agree to use at least one highly effective method of contraception throughout the study.

Exclusion Criteria:

Ocular conditions:

1. Any ocular condition in the study eye that in the opinion of the investigator would prevent improvement in visual acuity.
2. Proliferative diabetic retinopathy in the study eye.
3. History of panretinal scatter photocoagulation(PRP)in the study eye within 4 months prior to screening, and/or anticipated need for PRP in the 3 months following randomization.
4. Active optic disc or retinal neovascularization, rubeosis iridis, active or history of choroidal neovascularization in the study eye.
5. History of pars plana vitrectomy at any time, intraocular surgery in the study eye within 90 days prior to screening.
6. History of use of intravitreal injectable or periocular depots corticosteroids (other than triamcinolone acetonide)within 3 months prior to the screening visit in the study eye.
7. Patients who have previously received triamcinolone acetonide in the study eye:

   * The intended dose for each triamcinolone acetonide injection was more than 4 mg.
   * The most recent dose was less than 3 months prior to the screening visit.
   * Any treatment-related adverse event that was seen, and in the opinion of the investigator, has the potential to worsen or reoccur with study treatment.
8. Patients who have previously received anti-VEGF therapy within 3 months prior to the screening visit in the study eye.
9. Uncontrolled glaucoma or glaucoma treated by 2 or more medications.
10. Aphakia or intraocular lens placement in the anterior chamber of the study eye.
11. Any active ocular infection; any history of recurrent or chronic infection or inflammation in the study eye.
12. History of herpetic infection in either eye.
13. History of corneal pathology/surgery
14. Contact lens use at any time during the study.

    Systemic conditions:
15. Uncontrolled systemic disease.
16. Poorly controlled diabetes mellitus.
17. Impaired renal function
18. Poorly controlled arterial hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
change from baseline of central retinal thickness as determined by logOCT | Week 12

SECONDARY OUTCOMES:
Proportion of patients with an improvement in best corrected visual acuity (BCVA) | Week 12
Change in macular volume and retinal thickness from baseline to Week 12 and Week 24 | Baseline, Week 12, Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Massin, MD, Study Chair — Lariboisière Hospital, Paris
Locations (65):
- United States (14):
  - Center 1115, Phoenix, Arizona
  - Center 1116, Phoenix, Arizona
  - Center 1108, Fort Myers, Florida
  - Center 1106, Chicago, Illinois
  - Center 1105, Indianapolis, Indiana
  - Center 1101, Boston, Massachusetts
  - Center 1109, Boston, Massachusetts
  - Center 1111, Boston, Massachusetts
  - Center 1114, Traverse, Michigan
  - Center 1112, Toms River, New Jersey
  - Center 1107, Lynbrook, New York
  - Center 1110, Pittburgh, Pennsylvania
  - Center 1104, Nashville, Tennessee
  - Center 1103, San Antonio, Texas
- Australia (4):
  - Center 2003, Chatswood
  - Center 2002, Melbourne
  - Center 2004, Murdoch
  - Center 2001, Sydney
- Belgium (3):
  - Center 1302, Antwerp
  - Center 1301, Brussels
  - Center 1303, Wilrijk
- Czechia (6):
  - Center 1704, Brno
  - Center 1701, Hradec Králové
  - Center 1703, Ostrava
  - Center 1702, Prague
  - Center 1705, Prague
  - Center 1706, Zlín
- France (5):
  - Center 1401, Dijon
  - Center 1402, Marseille
  - Center 1405, Nantes
  - Center 1403, Paris
  - Center 1404, Paris
- Germany (7):
  - Center 1504, Ahaus
  - Center 1502, Darmstadt
  - Center 1503, Freiburg im Breisgau
  - Center 1501, Karlsruhe
  - Center 1506, Leipzig
  - Center 1507, Münster
  - Center 1505, Saarbrücken
- Israel (9):
  - Center 1907, Afula
  - Center 1906, Beer Yakov
  - Center 1909, Beersheba
  - Center 1903, Jerusalem
  - Center 1908, Kfar Saba
  - Center 1902, Petah Tikva
  - Center 1901, Rehovot
  - Center 1904, Tel Aviv
  - Center 1905, Tel Litwinsky
- Italy (7):
  - Center 1604, Florence
  - Center 1601, Milan
  - Center 1607, Milan
  - Center 1610, Rome
  - Center 1606, Saronno
  - Center 1608, Udine
  - Center 1609, Verona
- Poland (2):
  - Center1801, Bydgoszcz
  - Center 1802, Gdansk
- Spain (8):
  - Center 1205, Alicante
  - Center 1201, Barcelona
  - Center 1202, Barcelona
  - Center 1204, Oviedo
  - Center 1206, Santiago de Compostela
  - Center 1208, Seville
  - Center 1209, Valencia
  - Center 1203, Valladolid